CLINICAL TRIAL: NCT06500689
Title: Efficacy and Safety of Allisartan Isoproxil/Sustained-Release Indapamide in Patients With Essential Hypertension Uncontrolled With Allisartan Isoproxil: A Phase III, Multicenter, Randomized, Double-blind, Parallel-controlled, 52-week Clinical Study
Brief Title: To Assess Allisartan Isoproxil/Sustained-Release Indapamide in Patients With Essential Hypertension Uncontrolled With Allisartan Isoproxil
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAL0108A103
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Essential Hypertension
Keywords: Allisartan isoproxil; Indapamide; Essential hypertension; Systolic BP; Diastolic BP
MeSH Terms: conditions — Essential Hypertension | interventions — allisartan isoproxil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allisartan Isoproxil/Sustained-Release Indapamide Group (Experimental): Patients will be treated with one Allisartan Isoproxil/Sustained-Release Indapamide (240 mg/1.5 mg) tablet and one placebo of Allisartan Isoproxil during the double-blind period (Week 1~Week 12) and one Allisartan Isoproxil/Sustained-Release Indapamide (240 mg/1.5 mg) tablet during the open-label period (Week 13~Week 52) once daily.
  Interventions: Drug: Allisartan Isoproxil/Sustained-Release Indapamide
- Allisartan Isoproxil Group (Active Comparator): Patients will be treated with one Allisartan Isoproxil (240 mg) and one placebo of Allisartan Isoproxil/Sustained-Release Indapamide (240 mg/1.5 mg) tablet during the double-blind period (Week 1~Week 12) and one Allisartan Isoproxil/Sustained-Release Indapamide (240 mg/1.5 mg) tablet during the open-label period (Week 13~Week 52) once daily.
  Interventions: Drug: Allisartan Isoproxil

INTERVENTIONS:
Drug: Allisartan Isoproxil/Sustained-Release Indapamide — Double-blind period (Week 1~Week 12): Allisartan Isoproxil/Sustained-Release Indapamide.
  Open-label period (Week 13~Week 52): Allisartan Isoproxil/Sustained-Release Indapamide.
  Arms: Allisartan Isoproxil/Sustained-Release Indapamide Group
Drug: Allisartan Isoproxil — Double-blind period (Week 1~Week 12): Allisartan Isoproxil.
  Open-label period (Week 13~Week 52): Allisartan Isoproxil/Sustained-Release Indapamide.
  Arms: Allisartan Isoproxil Group

SUMMARY:
The main objective of the study will be to assess the efficacy and safety of Allisartan Isoproxil/sustained-release indapamide (240 mg/1.5 mg) in patients with mild to moderate essential hypertension uncontrolled after 4-week treatment with Allisartan Isoproxil (240 mg).

DETAILED DESCRIPTION:
Allisartan isoproxil is a novel angiotensin receptor blocke available in China for over ten years and has the same active compound EXP3174 with losartan, while sustained-release indapamide is a long-standing thiazide-type diuretic. The novel single-pill combination of allisartan isoproxil and sustained-release indapamide exerts synergistic antihypertensive effects.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients 18-75 years old with mild to moderate essential hypertension;
2. Patients who meet one of the following criteria when screening:

   1. Untreated patients (either newly diagnosed essential hypertension or those patients with a history of hypertension but have not been taking any antihypertensive drugs for at least 2 weeks before the first visit) must have an office msSBP ≥ 150 mmHg and < 180 mmHg and msDBP<110 mmHg;
   2. Patients who had not received regular treatment with allisartan isoproxil (240 mg/day) (less than 4 weeks of medication intake or a history of missing doses for 5 or more days within the 4 weeks before screening) with the msSBP of 140 mmHg≤ SBP <180 mmHg and DBP<110 mmHg;
   3. Patients currently receiving other antihypertensive agents (non-study medications for at least 2 weeks prior to screening) with the msSBP of 140 mmHg≤ SBP <180 mmHg and DBP<110 mmHg, and the clinician determined that it was appropriate to switch to allisartan isoproxil (240 mg/day);
   4. Patients who have been stably treated with allisartan isoproxil (240 mg/day) for at least 4 weeks with the msSBP of 140 mmHg≤ SBP <180 mmHg and DBP<110 mmHg.
3. During randomization for the double-blind treatment period, msSBP should be 140 mmHg≤ SBP <180 mmHg and DBP<110 mmHg;
4. Participants enrolled in the ABPM study should have 24-hour mean ambulatory blood pressure ≥130/80 mmHg after 4 weeks of monotherapy treatment;
5. Patients who understand and sign the informed consent form.

Key Exclusion Criteria:

1. Patients with secondary hypertension;
2. Patients with msSBP ≥180 m mHg and/or msDBP≥110 mmHg, or withhypertensive emergency or hypertensive urgency.
3. Patients who have taken three or more antihypertensive drugs (including single-pill combination) simultaneously within one month prior to screening.
4. Patients with history of heart failure (New York Heart Association (NYHA) Functional Classification class III and IV), acute coronary syndrome, percutaneous coronary intervention, or other serious heart diseases (such as cardiogenic shock, moderate or severe heart valvular disorders, atrioventricular block second or third degree, bradycardia (with a heart rate <50 beats per minute), severe arrhythmias) in the past 6 months.
5. Patients with history of severe cerebrovascular diseases (such as hypertensive encephalopathy, cerebrovascular injury, stroke, transient ischemic attack) in the past 6 months.
6. Patients with aortic aneurysm, aortic dissection, or dissecting aneurysm.
7. Patients with severe renal insufficiency (Cr>1.5 times the upper limit of normal).
8. Patients with hypokalemia or hyperkalemia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean seated systolic blood pressure (msSBP) after 12 weeks of randomized, double-blind treatment | week 1, week 12.

SECONDARY OUTCOMES:
Change from baseline in mean seated systolic blood pressure (msSBP) after 4 and 8 weeks of randomized, double-blind treatment | week 1, week 4, week 8.
Change from baseline in mean seated diastolic blood pressure (msDBP) after 4, 8, and 12 weeks of randomized, double-blind treatment | week 1, week 4, week 8, week 12.
The proportion of responders to antihypertensive treatment after 12 weeks of randomized, double-blind treatment. (Responders are the participants achieving SBP/DBP<140/90 mmHg or a reduction from baseline of >20 mmHg in msSBP and/or >10 mmHg in msDBP. ) | week 1, week 12.
The proportion of patients meeting the mean sitting blood pressure target (SBP/DBP <140/90mmHg) after 4, 8, and 12 weeks of randomized, double-blind treatment | week 1, week 4, week 8, week 12.
The proportion of patients with the mean sitting blood pressure SBP/DBP <130/80mmHg) after 4, 8, and 12 weeks of randomized, double-blind treatment | week 1, week 4, week 8, week 12.
Change from baseline in msSBP after 20, 28, 40, and 52 weeks of treatment | week 1, week 20, week 28, week 40, week 52.
Change from baseline in msDBP after 20, 28, 40, and 52 weeks of treatment | week 1, week 20, week 28, week 40, week 52.
The proportion of patients meeting the mean sitting blood pressure target (SBP/DBP <140/90mmHg) after 52 weeks of treatment | week 1, week 52.
The proportion of patients with the mean sitting blood pressure SBP/DBP <130/80mmHg) after 52 weeks of treatment | week 1, week 52.

OTHER OUTCOMES:
Change from baseline in 24-hour mean systolic and diastolic blood pressure during ambulatory blood pressure monitoring (ABPM) after 12 weeks of randomized, double-blind treatment | week 1, week 12.
Change from baseline in daytime mean systolic and diastolic blood pressure during ambulatory blood pressure monitoring (ABPM) after 12 weeks of randomized, double-blind treatment | week 1, week 12.
Change from baseline in nighttime mean systolic and diastolic blood pressure during ambulatory blood pressure monitoring (ABPM) after 12 weeks of randomized, double-blind treatment | week 1, week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Jinxiu Lin, MD, Principal Investigator — The First Affiliated Hospital of Fujian Medical University, Fuzhou 350212, China
Locations (40):
- China (40):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Xuancheng People's Hospital, Xuancheng, Anhui
  - Aerospace Central Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Chongqing University Affiliated Three Gorges Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Gansu Provincial People's Hospital, Lanzhou, Gansu
  - Shunde Hospital of Southern Medical University, Foshan, Guangdong
  - Guangdong Medical University Affiliated Hospital, Zhanjiang, Guangdong
  - Nanning First People's Hospital, Nanning, Guangxi
  - Hebei Provincial People's Hospital, Shijiazhuang, Hebei
  - Shijiazhuang People's Hospital, Shijiazhuang, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Daqing People's Hospital, Daqing, Heilongjiang
  - Kaifeng Traditional Chinese Medicine Hospital, Kaifeng, Henan
  - Chinese Medicine Dongfeng General Hospital, Shiyan, Hubei
  - Wuhan First Hospital, Wuhan, Hubei
  - Wuhan Fourth Hospital, Wuhan, Hubei
  - Wuhan Sixth Hospital, Wuhan, Hubei
  - Xiangya Second Hospital of Central South University, Changsha, Hunan
  - Yueyang Central Hospital, Yueyang, Hunan
  - Yueyang People's Hospital, Yueyang, Hunan
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - The First Affiliated Hospital of Gannan Medical College, Ganzhou, Jiangxi
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Tonghua Central Hospital, Tonghua, Jilin
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Nanchong Central Hospital, Nanchong, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Li Huili Hospital of Ningbo Medical Center, Ningbo, Zhejiang
  - Quzhou People's Hospital, Quzhou, Zhejiang
  - Wenzhou Medical University Affiliated First Hospital, Wenzhou, Zhejiang